CLINICAL TRIAL: NCT01540656
Title: Mechanical Nerve Stimulation in the Treatment of Post Prostatectomy Incontinence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2011-118
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Urinary Incontinence; Radical Prostatectomy
Keywords: Stress incontinence; Incontinence; prostate cancer; Radical Prostatectomy vibration; nerve stimulation
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): This group will receive immediate TMNS treatment beginning at baseline and ending at the 6 week point of the study.
  Interventions: Device: Transcutaneous mechanical nerve stimulation (TMNS) (FERTI CARE)
- Group 2 (Active Comparator): This group will receive delayed TMNS treatment beginning at the 6 week point of the study and ending at 12 weeks.
  Interventions: Device: Transcutaneous mechanical nerve stimulation (TMNS) (FERTI CARE)

INTERVENTIONS:
Device: Transcutaneous mechanical nerve stimulation (TMNS) (FERTI CARE) — A medical vibrator (FERTI CARE personal, Multicept A/S, Albertslund, Denmark) will be used. The stimulation works through a vibrating disc of hard plastic with a diameter of 3.5 cm. The stimulation point will be the frenulum of the glans penis. The stimulation will be performed with a vibration amplitude of 2 mm and a frequency of 100 Hz.
  A daily stimulation sequence consisting of 10 seconds of stimulation followed by a 10 second pause repeated 10 times will be used through 6 weeks.
  Other Names: FERTI CARE personel, Multicept A/S, Albertslund, Danmark; TMNS

SUMMARY:
During transcutaneous mechanical nerve stimulation in spinal cord injured men an increase in pressure was observed in the external urethral sphincter along with an increase in bladder capacity. In a subsequent study it was demonstrated that Transcutaneous Mechanical Nerve Stimulation (TMNS) in women could induce pressure increment of the external urethral sphincter. A pilot study have since shown that after 6 weeks of stimulation 24 out of 33 women suffering from urinary stress incontinence were able to contract their pelvic floor muscles and had become free of symptoms. Another pilot study has shown promising effect on the overactive bladder syndrome. Furthermore pilot studies in men who are incontinent after a radical prostatectomy have shown promising results. A randomized investigation of TMNS applied in the immediate period after a radical prostatectomy to investigate effects on both continence and erectile function is on going.

The present study aims to treat urinary incontinence in men who are still incontinent more than 1 year after a radical prostatectomy. A medical vibrator is used daily for a period of 6 weeks and the results of the treatment is then evaluated. The participants will be randomized to 2 groups. Group 1 starts vibration treatment at base line and group 2 starts after 6 weeks when group 1 is done. The groups are compared at baseline, at 6 weeks and at 12 weeks.

The stimulation will be performed at the frenulum of the glans penis every day for 6 weeks with an amplitude of 2 mm and a frequency of 100 Hz. Results will be evaluated on the basis of questionnaires, micturition diaries and diaper tests.

If the investigators are able to demonstrate a significant reduction in the incontinence symptoms in the subjects the investigators asses that vibration can be a way of reestablishing normal continence in men after a radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Men who have undergone a radical prostatectomy at least 1 year prior to enrollment
* Incontinence induced by the surgery (at least 8 g/24 hours)
* Capable of understanding study information and following treatment

Exclusion Criteria:

* Incontinence before radical prostatectomy
* Treatment with anticholinergic medications
* Radiation or hormone treatment
* Previous surgical treatment of incontinence
* Acute illness (including infection, trauma and haematuria)
* Faecal incontinence
* Known neurological disease
* Known Bladder pathology on cystoscopy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
24 hour Diaper test (weight in grams) at 6 weeks | Assessment at baseline and again after 6 weeks
  Participants will be provided diapers and they will wear them for 24 hours. The weight of all used diapers is then measured to assess how much urine is leaking.
  The main outcome measure is the difference in leakage between groups 1 and 2 at 6 weeks (when group 1 has received treatment and group 2 has not).

SECONDARY OUTCOMES:
24 hour Diaper test (weight in grams) at 12 weeks | Assessment at baseline and again after 12 weeks
  Participants will be provided diapers and they will wear them for 24 hours. The weight of all used diapers is then measured to asses how much urine is leaking.
  Here the leakage between groups 1 and 2 is measured at 12 weeks (when both groups have received treatment ).
Micturition diary | Assessment at baseline after 6 weeks and again after 12 weeks
  The number of involuntary incontinence and normal micturition episodes are evaluated based on a patient diary. Here the difference in number of incontinence episodes between groups 1 and 2 are calculated at 6 weeks (when only group 1 has received treatment) and at 12 weeks (when both groups have received treatment).
Validated symptom score (ICI-Q) | Assessment at baseline after 6 weeks and again after 12 weeks
  The ICI-Q symptom score includes changes in incontinence and micturition patterns and patients' subjective assessment of their symptoms.
  The scores are evaluated and differences between groups 1 and 2 are calculated at 6 weeks (when only group 1 has received treatment) and at 12 weeks (when both groups have received treatment).
International Prostate symptom score (I-PSS)questionnaire | Assessment at baseline after 6 weeks and again after 12 weeks
  The total score as well as storage and voiding domains are evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Fode, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Department of Urology, Herlev Hospital, Herlev

REFERENCES:
- [Derived] Fode M, Sonksen J. Penile vibratory stimulation in the treatment of post-prostatectomy incontinence: a randomized pilot study. Neurourol Urodyn. 2015 Feb;34(2):117-22. doi: 10.1002/nau.22536. Epub 2013 Nov 27. PMID 24285576